CLINICAL TRIAL: NCT02851875
Title: Duke Scleroderma Clinic Patient Registry
Status: Terminated | Type: Observational
Why Stopped: Low enrollment and no plans for analysis
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00067280
Record Dates: First submitted 2016-04-18; First posted 2016-08-02 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2020-09

CONDITIONS: Scleroderma; Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic | interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Registry

SUMMARY:
The purpose of the Duke Scleroderma Registry (DSScR) is to obtain information about scleroderma. This information could be used in future research to increase the understanding of disease mechanisms, treatments, and outcomes. This research may also help develop new therapies, novel measures of disease assessment or identify previously unknown manifestations of the diseases. A prospectively followed cohort is an integral component of future translational and clinical research programs. A registry for scleroderma would allow for information to be gleaned about patients in "real-world situations" in an effort to improve the reality, generalizability and applicability of information gathered.

DETAILED DESCRIPTION:
The Duke Scleroderma Registry (DSScR) will include 3 types of data collected at each standard of care office visit, generally every 3-6 months. The data will include:

1. Clinical data obtained by clinicians and entered electronically into a secure database
2. Laboratory, procedure, and imaging data obtained over the course of clinical care
3. Photographs of clinically relevant physical findings.

Data that will be stored include historical data on patients' disease and concurrent medical conditions, physical exam findings, laboratory values, imaging and other diagnostic testing results, detailed list of medications and treatments, and quality of life questionnaire data. Historical information will include detailed medical, obstetric, surgical, procedural, social, and family history of disease comparable to information gathered at a typical initial visit. No protected health information will be collected or stored on family members. Data collected will be stored in a secure computer database as well as in a clinic note and will be used for patient care purposes. Protected health information (PHI) that will accompany subject data include name, medical record number, address, phone number, date of birth, dates of diagnoses, dates of procedures, and dates of clinic visits.

The database will be maintained indefinitely; there is no planned endpoint to the collection of the data and maintenance of the database as the investigators are planning a long term prospective evaluation of persons with these diseases.

Subjects will be serially approached/recruited from existing patients in the Duke Rheumatology Adult Clinic. The project will be introduced to each prospective subject by someone involved in their clinical care. A waiver of consent and Health Insurance Portability and Accountability Act (HIPAA) authorization has been filed for the Duke Scleroderma Registry. Persons who have been diagnosed with scleroderma will be identified through monitoring of outpatient clinic lists and the inpatient consult service.

Research records will be archived upon completion of the study. Subject initials and study number will be used to identify subjects in the research material and on research specimens. All electronic data is stored on the shared drive and secured through the following Duke Health Technology Services approved methods: access rights granted and terminated for authorized users only, secure laptops and workstations, individual identifier plus password protection, routine electronic back up, network restrictions.

During the initial screening process, no identifying information (e.g., name, address) will be kept. During the consent process, participants will be informed of data storage and confidentiality safeguards, which are practiced according to HIPAA regulations. Each participant will be assigned a unique identifier (ID) number. All data will be de-identified and coded with this number only.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of systemic sclerosis or Scleroderma as identified by the 2013 American College of Rheumatology classification criteria

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 and older with a history of scleroderma or systemic sclerosis.
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2016-04; Primary Completion 2018-05-07 (Actual); Study Completion 2018-05-07 (Actual)

PRIMARY OUTCOMES:
Change in disease activity as measured by Rodnan Skin Score | Change from baseline at 10 years
  The Rodnan skin score is a discrete measure of skin thickness that can change through time and in response to medication.
Change in disease activity as measured by patient reported Scleroderma Health Associated Questionnaire (SHAQ) | Change from baseline at 10 years
  The SHAQ is a measure of health and disability that produces a discrete value that can change through time and in response to medication.

CONTACTS AND LOCATIONS:
Overall Officials: Ankoor Shah, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No